CLINICAL TRIAL: NCT04618679
Title: Application of 18F-FDOPA PET in Research of the Association Between HCV Infection and Parkinson's Disease.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201912133MIND
Record Dates: First submitted 2020-11-01; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-10

CONDITIONS: Hepatitis C
Keywords: HBV,Parkinson's disease,18F-FDOPA PET
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 18F-FDOPA PET: Patients with HCV infection receive 18F-FDOPA PET to investigate preclinical Parkinson's disease.

SUMMARY:
-[18F]Fluoro-L-3,4-dihydroxyphenylalanine (18F-FDOPA) positron emission tomography (PET) is a imaging marker for presynaptic dopaminergic neuronal function. The decreased uptake of 18F-FDOPA in the posterior putamen is demonstrated in the early course of PD, and could differentiate early PD from healthy controls. The objective of this study is to investigate the evidence of presynaptic dopaminergic neuronal dysfunction in the preclinical stage of PD, which may be associated with HCV infection.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second-most neurodegenerative disease in Taiwan. It is characterized by the progressive loss of dopaminergic neurons in the substantia nigra pars compacta (SNpc). The estimated incidence of PD ranging from 10-18 per 100,000 person-years with a tread of increasing number over past decades. Although the exact mechanisms of PD have not yet fully clear, many pathological process have shown to be involved in the pathogenesis like abnormal alpha-synuclein, activation of microglia and astrocyte, mitochondrial dysfunction, oxidative stress, and so on.

Several characteristics have been considered to increase the risk of having PD. Epidemiologic studies have suggested that patients with HCV infection might have higher risk of PD. It is common that patients with chronic HCV infection manifest with central nervous system manifestations, such as depression, fatigue, and cognitive dysfunction. A previous epidemiologic study in Taiwan with a total of 62,276 subjects showed that there is significant correlation between PD and hepatitic C virus (HCV) infection. In the study, the crude odds ratio for having PD was 1.94 for HCV patients.

HCV is positive-stranded RNA virus of Flaviviridae family. Flaviviridae family has many viruses demonstrating neurotropic character and may be associated with encephalopathy. Decreased monoamine transporter binding activity had also been found in HCV infected patients who had symptoms of chronic fatigue and cognitive impairment. HCV can cross blood-brain barrier and has the ability to replicate in the central nervous system. Animal study has shown that HCV infection may up-regulate the inflammatory cytokines, such as sICAM-1, LIX, and RANTES, in the rat midbrain neuron-glia coculture and induced dopaminergic neuronal toxicity. The elevation of choline/creatine ratio on proton magnetic-resonance spectroscopy is also indicative of inflammatory status of brain in patients with chronic HCV infection. it is possible that the direct infection of HCV into the brain induce inflammatory status by microglia/macrophages and contribute to subsequent neurodegeneration. Chronic HCV infection is also associated with systemic cytokine activation including interferon-α and tumor necrosis factor α, which may also affect the neuronal function. It has been reported that the viral eradication on the patients infected by HCV had change of neurocognitive function.

6-[18F]Fluoro-L-3,4-dihydroxyphenylalanine (18F-FDOPA) is an analog of L-dihydroxyphenylalanine (L-DOPA), which is the precursor of dopamine. L-DOPA is carried into the brain through neutral amino acid transport system and converted to domapine by aromatic L-amino acid decarboxylase (AADC) in dopaminergic neurons. Use 18F-FDOPA as a tracer of positron emission tomography (PET) imaging, the dopamine synthesis rate and presynaptic dopaminergic neuronal function can be reflected by the uptake of 18F-FDOPA in dopaminergic neurons. The decline of 18F-FDOPA is indicative of dopaminergic neurons dysfunction and can be used as imaging marker of the severity of PD. The posterior putamen receives the dopaminergic projections from the ventrolateral part of the substantia nigra and is affected earliest in the disease course of PD. 18F-FDOPA has been shown its capacity in differentiating early PD and healthy controls in previous study with lower metabolism in the dorsal putamen even in the early course of PD.

In this project, 18F-FDOPA PET is used as an imaging marker of striatal dopaminergic dysfunction in patients with HCV infection. We will try to detect the subclinical and preclinical stages of parkinsonism for these patients.

ELIGIBILITY:
Adults (older than 20-year-old) with HCV infection and agree to accept 18F-FDOPA PET examination.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient department of hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-11-02 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Application of 18F-FDOPA PET in research of the association between HCV infection and Parkinson's disease. | 2 weeks
  To evaluate the uptake of 18F-FDOPA in the basal ganglia of patients with HCV infection. Use 18F-FDOPA PET as an imaging marker to diagnosis preclincal Parkinson's disease in patients with HCV infection.

SECONDARY OUTCOMES:
Application of 18F-FDOPA PET in research of the association between HCV infection and Parkinson's disease. | 2 weeks
  To compare the findings of 18F-FDOPA PET with the disease status of HCV infection and investigate possible correlation between the severity of Parkinson's disease and HCV infection status.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ju v Liu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Douliu, Yunlin County, Taiwan